CLINICAL TRIAL: NCT02933177
Title: Study on Effectiveness of Flash Mediation Therapy in the Context of Acute Psychological and Behavioral Symptoms of Dementia in Nursing Homes
Brief Title: Effectiveness of Flash Mediation Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 69HCL16_0442
Record Dates: First submitted 2016-10-12; First posted 2016-10-14 (Estimated); Last update posted 2017-12-02 (Actual); Status verified 2017-08

CONDITIONS: Dementia
Keywords: Dementia; Alzheimer disease; Behavioral and Psychological Symptoms of Dementia; non-drug intervention
MeSH Terms: conditions — Dementia; Alzheimer Disease; Behavior

ARMS (2):
- 2 months control condition - 4 months chariot-flash (Experimental): 200 patient , in 15 nursing homes randomly will be exposed two months in the control condition (usual intervention) and 4 months in the experimental condition (chariot-flash intervention). The experimental condition is to propose the "chariot-flash" in emergency during the emergence or increase of productive symptoms.
  Interventions: Behavioral: 2 months control condition - 4 months chariot-flash
- 4 months control condition-2 months chariot flash (Experimental): 200 patient, in 14 other nursing homes will be exposed 4 months in the control condition and 2 months in the experimental condition
  Interventions: Behavioral: 4 months control condition-2 months chariot flash

INTERVENTIONS:
Behavioral: 2 months control condition - 4 months chariot-flash — The control condition is to propose the usual procedures for the management of productive symptoms during the emergence or increase of these symptoms.
  The "chariot-flash" condition is a chariot with eleven drawers. Each drawer contains an activity (lasting about 15 minutes):
  * Boards of known photographs to recall autobiographical memories
  * Newspapers to read, talk, associate memories around an article
  * Massage Oil, refreshing wipes, cream to reconnect with the body
  * Clay, cookie pieces, washable felt and paper to create shapes, draw.
  * Walk with a person of the healthcare team the case of behavioral disorders in type of ambulation and untimely exit .
  * Listening to music
  * Relaxation-Breathing
  * Cushion, foam balls to vent his energy on secure hardware.
  * Plush doll or to invest a vector object of affection and empathy
  * Sensory flash balls that the patient can squeeze, throw, roll.
  * Games with which the patient can play according to its possibilities.
  Arms: 2 months control condition - 4 months chariot-flash
Behavioral: 4 months control condition-2 months chariot flash — The control condition is to propose the usual procedures for the management of productive symptoms during the emergence or increase of these symptoms.
  The "chariot-flash" condition is a chariot with eleven drawers. Each drawer contains an activity (lasting about 15 minutes):
  * Boards of known photographs to recall autobiographical memories
  * Newspapers to read, talk, associate memories around an article
  * Massage Oil, refreshing wipes, cream to reconnect with the body
  * Clay, cookie pieces, washable felt and paper to create shapes, draw.
  * Walk with a person of the healthcare team the case of behavioral disorders in type of ambulation and untimely exit .
  * Listening to music
  * Relaxation-Breathing
  * Cushion, foam balls to vent his energy on secure hardware.
  * Plush doll or to invest a vector object of affection and empathy
  * Sensory flash balls that the patient can squeeze, throw, roll.
  * Games with which the patient can play according to its possibilities.
  Arms: 4 months control condition-2 months chariot flash

SUMMARY:
In order to offer a non-drug intervention for caregivers in nursing home to respond promptly to a behavioral crisis with an appropriate response to each patient, a chariot has been developed by the Institute of Ageing Well Korian (Institut du Bien Vieillir Korian) to bring together eleven mediation activities. These activities lasting about 15 minutes are based on emotion (reminiscent, games) and sensory interventions (music, massage, touch) to decentralize patient stimulus that disturbs and focus on a subject not disruptive. This emergency intervention should provide a reduction in Behavioral and Psychological Symptom of Dementia (BPSD) of nursing home patients. The main objective is to measure its immediate effect on productive symptoms (agitation, aberrant motor behavior and disinhibition). The secondary objectives are to measure its immediate impact on the well-being and psychotropic treatments, and measure its effect after two months and after four months on all BPSD with a focus on agitation, the administration of psychotropic drugs, the hospitalizations and the number of falls.

ELIGIBILITY:
Inclusion Criteria:

* People ability to object and does not oppose either by themselves or through a trusted person referred to in Article L. 1111-6 of the Code of Public Health, failing thereof, by the family, or, if a person talking to the person close and stable ties. For adults under guardianship, permission must be given by the legal representative of the person. The research will benefit from the backing of Persons Protection Committee (PPC) prior to its implementation;
* Man or woman over 60 years;
* patient living in one of the nursing homes participating in the project;
* Patient completing the diagnostic criteria for major neurocognitive disorder according to Diagnostic and Statistical Manual of Mental Disorders V criteria (DSM-V)
* The patient must have at least one of these productive symptoms (agitation, aberrant motor behavior, disinhibition) listed by the NPI-NH (score> 2 at least one of these items)

Exclusion Criteria:

* Deafness or blindness may compromise patient assessment or participation in the intervention

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 241 (Actual)
Dates: Start 2016-05; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Change in number of disorders | until 4 months
  the number of disorders are evaluated with Cohen Mansfield Agitation Inventory (CMAI) before and 30 minutes after each intervention.
  The original version of the CMAI is initially planned to study the frequency of these disorders. However, the goal being to study the decrease in productive symptoms, after using the "chariot-flash", only the number of this item will be considered (between 0 and 29). For example in this modified version, for the item "pace, aimless wandering" nursing team can answer "present" or "absent" instead of (never, less than once a week, once or twice per week, a few times over week, one to two times daily, several times a day, several times per hour)

SECONDARY OUTCOMES:
Change in score of well-being | until 4 months
  the score of well-being is assessed using the Instant Well-Being scale (Evaluation Instantané du Bien-Etre : EVIBE) before and 30 minutes after each intervention .
  The EVIBE is a visual analogue scale for reporting the status of well-being of the patient at a specific time. On a graduated scale from 0 to 5, the caregiver should position a cursor position to the left corresponding to the feeling of well-being the lowest and the right position to the feeling of well-being the highest.
change in psychotropic drugs prescribed | until 4 months
  The caregiver or doctor will check on a board what are the treatments that have been added or modified (compared to the usual treatment) in response to behavioral disorder
change in score of BPSD | before the beginning of the study, at 2 months, 4 months and 6 months
  the score of BPSD is assessed using the neuropsychiatric inventory nursing home version (NPI-NH).
  Each of the 12 BPSD (delusions, hallucinations, agitation, depression, anxiety, excitement, apathy, disinhibition, depression, motor aberrant behavior, sleep and appetite) is evaluated on 12 depending on its frequency and severity (global score =144).
change in level of agitation | before the beginning of the study, at 2 months, 4 months and 6 months
  the level of agitation is assessed using the original version of CMAI. The CMAI lists 29 agitation and aggressive behaviors by frequency (0: not evaluable 1: never, 2: less than once a week 3 : once or twice per week, 4 : a few times over week, 5: one to two times daily, 6 : several times a day, 7 : several times per hour) to obtain a score ranging from 0-203.
change in the number of administered psychotropic drugs. | before the beginning of the study, at 2 months, 4 months and 6 months
  The caregiver or doctor will check on a board on which is written all psychotropic treatments that the patient takes and the dosage
The number of hospitalization | at 2 months, 4 months and 6 months
  The caregiver or doctor will refer in a table the different hospitalizations during the study and their date
The number of fall | at 2 months, 4 months and 6 months
  The caregiver or doctor will refer in a table the different falls during the study and their date.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Krolak Salmon, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hôpital des Charpennes Centre de Recherche Clinique "Vieillissement-Cerveau-Fragilité", Lyon, France

IPD SHARING:
Plan to Share IPD: No